CLINICAL TRIAL: NCT05773768
Title: EHRA-PATHS: Addressing Multimorbidity in Elderly Atrial Fibrillation Patients Through Interdisciplinary, Patient-centred Systematic Care Pathways - Clinical and Health Economic Evaluation of New Care Pathways
Brief Title: EHRA-PATHS: Clinical and Health Economic Evaluation of New Care Pathways
Acronym: EHRA-PATHS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: EHRA-PATHS
Record Dates: First submitted 2023-02-15; First posted 2023-03-17 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- New care program (Experimental): The health care provider will use the EHRA-PATHS' newly developed care pathways to assess whether there is an indication for presence of risk factors and comorbidities. If this is the case, the care pathways will show possible next steps for confirming the presence of these risk factors and comorbidities. If confirmed, treatment according to the current guidelines should be initiated. Since this leads to an individualized management plan, procedures can differ between patients and will also depend on local processes.
  Interventions: Device: EHRA-PATHS software tool
- Routine clinical care (No Intervention): The health care provider follows current clinical practice with regards to history taking, physical examination etc.

INTERVENTIONS:
Device: EHRA-PATHS software tool — Newly developed care pathways integrated into a care-management software tool
  Arms: New care program

SUMMARY:
In elderly atrial fibrillation (AF) patients, AF is usually a manifestation of risk factors and comorbidities not only limited to cardiovascular diseases. Especially in elderly often more than two comorbidities are present. The presence of comorbidities also affects outcomes in AF patients. Current healthcare systems are single-disease focused, which increases the risk of underdiagnosing, replicating diagnostic tests and adverse drug-drug interactions, placing a high burden on healthcare costs. Healthcare systems and hospitals are in need of new care pathways to address the complexity of multimorbid AF patients and to reduce costs. The EHRA-PATHS consortium set out to address this need for change in management for multimorbid, elderly AF patients in Europe through the development of new care pathways. The aim of this study is to evaluate the current management of risk factors and comorbidities, and subsequently implement the newly developed care pathways and evaluate if these pathways lead to better management of risk factors and comorbidities in multimorbid, elderly AF patients, compared to current standard care.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed atrial fibrillation (paroxysmal, persistent or permanent)
* ≥65 years of age
* Willing and able to participate and to attend the scheduled follow-up visits.

Exclusion Criteria:

* Atrial fibrillation episode was due to a trigger (i.e. postoperative, infection, hyperthyroidism etc.)
* Life expectancy of less than 1 year
* Participation in another clinical study (registry studies not included)
* Severe cognitive impairment / dementia (defined based on MMSE and CDR scoring systems)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1300 (Estimated)
Dates: Start 2024-03-28 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Identification and management of risk factors and comorbidities | 6 months
  The number of risk factors and comorbidities that are identified and for which treatment is initiated during base mapping and at the end of the randomized controlled trial.

SECONDARY OUTCOMES:
AF symptom burden | 6 months
  Measured with the Atrial Fibrillation Severity Scale (AFSS) questionnaire
Quality of life (QoL) | 6 months
  Measured with the EuroQol five-dimensional five-level (EQ-5D-5L) questionnaire
Referrals to other disciplines | 6 months
  The referrals to other disciplines will consist of the number of referrals and the percentage of patients referred.
Patient and health care provider satisfaction | 6 months
  Measured with a patient and health care provider (HCP) satisfaction questionnaire
Healthcare resource use/costs | 6 months
  Measured with the iMedical Consumption Questionnaire (iMCQ)
HRQoL/utility | 6 months
  Measured with the EQ-5D-5L questionnaire (iMCQ)

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No